CLINICAL TRIAL: NCT04727918
Title: Comparison of Cold Biopsy Forceps vs Cold Snare for Diminutive Colorectal Polyp Removal: a Multicenter Randomized Controlled Trial
Brief Title: Comparison of Cold Biopsy Forceps vs Cold Snare for Diminutive Colorectal Polyp Removal
Acronym: BIOPANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriel RAHMI (Other)
Responsible Party: Sponsor-Investigator, Gabriel RAHMI, Principal Investagator, Medical Doctor, French Society of Digestive Endoscopy
Organization: French Society of Digestive Endoscopy (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFED 105
Record Dates: First submitted 2021-01-25; First posted 2021-01-27 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Polyps
Keywords: Polypectomy; Cold biopsy forceps; Cold snare polypectomy; Diminutive colorectal polyp

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold biopsy forceps (CBF) (Active Comparator): Patients will be allocated to the CBF arm after randomization (1:1)
  Interventions: Procedure: Polypectomy of diminutive colorectal polyps will be performed by CBF
- Cold snare polypectomy (CSP) (Active Comparator): Patients will be allocated to the CSP arm after randomization (1:1)
  Interventions: Procedure: Polypectomy of diminutive colorectal polyps will be performed by CSP

INTERVENTIONS:
Procedure: Polypectomy of diminutive colorectal polyps will be performed by CBF — All polypectomy procedures will be standardized amongst the study centers. Endoscopists with a minimal experience of at least 50 CBF and CSP performed the polypectomies CBF : The CBF will be performed using a standard biopsy forceps (Gluton Life ® Life Partners). Multiple biopsies bites were taken until complete resection (as many as needed).
  Arms: Cold biopsy forceps (CBF)
Procedure: Polypectomy of diminutive colorectal polyps will be performed by CSP — All polypectomy procedures will be standardized amongst the study centers. Endoscopists with a minimal experience of at least 50 CBF and CSP performed the polypectomies CSP : The CSB procedure will be performed using a 9 mm cold snare (Exacto ® Life Partners). One to two mm of normal surrounding mucosa will be ensnared around the base of the polyp, followed by mechanical excision without electrocautery
  Arms: Cold snare polypectomy (CSP)

SUMMARY:
European guidelines recommend the use of cold snare polypectomy (CSP) for removal of diminutive colorectal polyps (DCP)(5 mm or less). However, for DCP < 4 mm cold biopsy forceps (CBF) may be optional. Moreover, CBF remains the endoscopist's technique of choice for polyp resection and CSP is associated with a failure of specimen retrieval for histology in up to 6.8% of cases. In this study, the investigators aimed to compare the efficacy of CSP with CBF for removal of DCP in routine colonoscopy

ELIGIBILITY:
Inclusion Criteria:

* Routine colonoscopy
* Patient older than 18 years
* at least one polyp measuring ≤ 5 mm

Exclusion Criteria:

* inflammatory bowel disease
* polyposis syndrome, pregnancy
* inability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to compare CBF and CSP in terms of efficacy. The primary end-point is the rate of histological complete resection by anatomopathological examination. | through study completion, an average of 2 years.
  Complete histological resection was defined as the absence of visualized residual polyp after saline irrigation as well as negative biopsies of the polypectomy site

SECONDARY OUTCOMES:
Specimen retrieval rate (% time of polypectomy) | through study completion, an average of 2 years.
  specimen will be immediately suctioned into the operating channel.
Procedure time ( overall time between introduction and removal of colonoscope) | through study completion, an average of 2 years.
  measure of the time until complete polyp resection is obtained
Procedure related adverse events will be collected (adverse events : %, number of event for each groupe) during the procedure or during the follow up period (28 days). | All patients will be followed-up until 28 days post-colonoscopy.
  perforation, gastrointestinal and bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Georges Pompidou 20, rue Leblanc, Paris, France

REFERENCES:
- [Derived] Perrod G, Perez-Cuadrado-Robles E, Coron E, Pioche M, Becq A, Etchepare N, Danan D, Musquer N, Dray X, Laquiere A, Jais B, Broudin C, Benosman H, Cellier C, Rahmi G. Comparison of cold biopsy forceps vs cold snare for diminutive colorectal polyp removal: A multicenter non-inferiority randomized controlled trial. Clin Res Hepatol Gastroenterol. 2022 Mar;46(3):101867. doi: 10.1016/j.clinre.2022.101867. Epub 2022 Jan 14. PMID 35038578